CLINICAL TRIAL: NCT00467792
Title: Natural History of Urticaria Pigmentosa in Children
Acronym: UP
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Society for Pediatric Dermatology (Other)
Responsible Party: Sheila Galbraith, MD, Medical College of Wisconsin
Other Study IDs: UP
Record Dates: First submitted 2007-04-30; First posted 2007-05-01 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-12

CONDITIONS: Urticaria Pigmentosa
Keywords: urticaria pigmentosa; mastocytosis; mastocytomas
MeSH Terms: conditions — Urticaria Pigmentosa; Mastocytosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine how long the skin lesions usually last and what kind of symptoms and signs children with urticaria pigmentosa may develop over the years. This information will allow physicians to better care for patients who have been diagnosed with this disease and to provide their parents with more complete information regarding what to expect for the future of their child. This research is being done because many unanswered questions remain regarding children with urticaria pigmentosa and its course.

DETAILED DESCRIPTION:
This study involves children, of age 0-18 years old who are diagnosed with urticaria pigmentosa during their visit at the Pediatric Dermatology Clinic. Parents and child will be interviewed to gain medical and family history, in addition, the doctor will perform a physical exam and take a photograph. Children older than 4 years of age will complete the "Children Dermatology Life Quality Index." Children less than 4 years of age with an active disease will have laboratory tests requiring a sample of blood (1 teaspoon).

Patients will receive $50 for their first office visit as financial reimbursement for participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-18 years old at diagnosis of UP
* 3 or more mastocytomas (diagnosis can be based on clinical exam; biopsy only necessary if diagnosis is in question)
* patients recruited from Children's Hospital of Wisconsin Dermatology Clinic

Exclusion Criteria:

* Less than 3 mastocytomas
* Diffuse mastocytosis
* TMEP
* residence is out of Wisconsin/Illinois area or the United States

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study involves children, of age 0-18 years old who are diagnosed with urticaria pigmentosa during their visit at the Pediatric Dermatology Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Galbraith, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States